CLINICAL TRIAL: NCT02337075
Title: PAthway To Health (PATH): Fostering Culturally Appropriate Physical Activities Using Digital Technology in Indigenous Communities
Brief Title: PAthway To Health (PATH): Fostering Culturally Appropriate Physical Activities in Indigenous Communities
Acronym: PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Linda Li, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: H12-02526
Record Dates: First submitted 2015-01-05; First posted 2015-01-13 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: condition; preventing; physical activity
MeSH Terms: conditions — Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study used a delayed control design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Now Group - PATH Program (Experimental): The Now Group will receive the PATH program. They will participate in a brief education session, use a wearable physical activity tracker, and physical activity mentoring by an Activity Mentors. In Month 1 and 2, participants will meet with their Activity Mentor once every 2 weeks to review their physical activity status, activity goals, and the health programs available at the Centre. In Month 3 and 4, they will continue to use physical activity tracker but will no longer have regular meetings with the Activity Mentor.
  Interventions: Behavioral: PATH program; Device: Activity Mentor
- Later Group (Active Comparator): The Later Group will receive the PATH program in Month 1-2. Intervention will be provided two months later (i.e., Month 3 and 4).
  Interventions: Behavioral: PATH program; Device: Activity Mentor

INTERVENTIONS:
Behavioral: PATH program — A brief education session, use of a wearable physical activity tracker, and physical activity mentoring by an Activity Mentor every 2 weeks.
Device: Activity Mentor

SUMMARY:
Being physically active is important for everyone's health, but it is often challenging for people to start and sustain an activity routine. The investigators will develop and pilot test the PATH (PAthway To Health) program with Indigenous communities served by the Kwakiutl District Council (KDC) Health on North Vancouver Island. The project idea was conceived through a partnership between the communities and University of British Columbia health researchers. The PATH program will include an education sessions on how to be active, physical activity coaching by community health workers, and the use of Fitbit Flex (a wearable activity tracker). The investigators will develop a culturally appropriate online application to pair with Fitbit, which will provide instant feedback to individuals about their activity level. 60 community members will be recruited to test the PATH program. Their physical activity level, health status and use of activity resources at KDC Health Centres will be assessed.

DETAILED DESCRIPTION:
Background: Promoting an active lifestyle is a priority identified by the communities served by KDC Health. Statistics Canada estimates obesity in one in four adults based on 2007-2009 data, with higher prevalence among Indigenous people compared to non-Aboriginal population (between 26% and 36% among adults living off-reserve and on-reserve, respectively). Furthermore, Indigenous people also report higher prevalence of obesity associated complications, including diabetes, cardiovascular disease, and arthritis. The association between physical inactivity and obesity suggests that increasing physical activity is important.

KDC Health offers a variety of free programs to community members, however, the use of these services has been low. KDC Health has previously partnered with the CIHR-funded IMPAKT project, and has expressed a strong interest in developing an intervention to improve health and wellness in the communities.

Objectives:

1. To determine whether the PATH program can improve physical activity participation in the communities served by KDC Health.
2. To assess the effect of this program on reducing sedentary time, and increasing the use of health promotion and wellness services offered by KDC Health
3. To assess the correlation of physical activity levels and the secondary outcome measures among individuals who are living in the same household.

Methods: The investigators will conduct a community-based proof-of-concept randomized controlled trial (RCT) with 60 eligible participants. Only 1 member per household will be enrolled. If more than 1 member is interested, they will select 1 person by consensus or by a random draw.

After obtaining the baseline measures, participants will be randomly assigned to the 'Now Group' (target=30) or 'Later Group' (target=30).

The Now Group will participate in a brief education session held at the KDC Health Centre, use a wearable physical activity tracker (Fitbit Flex), and physical activity mentoring by a KDC Health Staff (the Activity Mentors). The Activity Mentors have received training for the project from the Principal Investigator. In Month 1-2, participants will meet with their Activity Mentor once every 2 weeks to review their physical activity status, activity goals, and the health programs available at the Centre. In Month 3-4, they will continue to use Fitbit Flex but will no longer have regular meetings with the Activity Mentor.

The Later Group will receive intervention two months later (i.e., Month 3-4).

The primary outcome measure will be the time spent in moderate/vigorous physical activity. In addition, time spent in sedentary behaviours will be recorded. Participants will wear a SenseWear Mini accelerometer for 7 days at baseline, 2 months, and 4 months. Secondary outcome measures include sedentary time measured with SenseWear Mini, health status that will be measured using the SF-36 (a generic measure of health-related quality of life), and body weight. Participants' use of KDC Health programs and their motivation to be physically active will also be recorded.

At the end of the program, participants will be interviewed for 30 minutes in person about their opinion on the intervention. Interviews will focus on 1) barriers/facilitators to being physically active, 2) their experience with the intervention, and 3) the nature of activities they engage in.

ELIGIBILITY:
Inclusion Criteria: Participants are eligible if they:

1. Are a person from KDC Health Member Nations
2. Are 19 years or older
3. Have no health condition that prevents them from being physically active
4. Are able to participate in a 4-month project -

Exclusion Criteria: Participants are not eligible to participate if they:

1. Do not meet the criteria above
2. Use medication that may impair activity tolerance (e.g., beta blockers),
3. Are unable to provide informed consent -

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Time spent in Moderate to Vigorous Physical Activity (MVPA), measured by SenseWear Mini accelerometer | Change from baseline in Time spent in MVPA at 2 months and 4 months
  Participants will wear a SenseWear Mini accelerometer for 7 days at baseline, and Months 2 and 4.

SECONDARY OUTCOMES:
Time spent in sedentary behaviours, measured by SenseWear Mini accelerometer | Change from baseline in time spent in sedentary behaviours at 2 months and 4 months
  Participants will wear a SenseWear Mini accelerometer for 7 days at baseline, and Months 2 and 4.
Change in Health Status, measured by SF-36 Questionnaire | Change from baseline health status at 2 months and 4 months
  SF-36 Questionnaire
Change in Body weight, measured by measured with a calibrated scale | Change from baseline body weight at 2 months and 4 months
  Measured with a calibrated scale

CONTACTS AND LOCATIONS:
Overall Officials: Linda Li, PT, PhD, Principal Investigator — Arthritis Research Canada
Locations (1):
- Arthritis Research Canada, Richmond, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No